CLINICAL TRIAL: NCT03250702
Title: Dar es Salaam Urban Cohort Hypertension Study
Brief Title: DUCS-DHD Determinants of Hypertension in Tanzania
Acronym: DUCS-HTN
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Goodarz Danaei, Associate Professor of Global Health, Harvard School of Public Health (HSPH)
Other Study IDs: IRB13-0852
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Hypertension; Obesity
Keywords: Tanzania; Observational; Sub-Saharan Africa; Treatment
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the Dar es Salaam Urban Cohort Hypertension Study (DUCS-HTN) was to determine the current prevalence, risk factors, and barriers to diagnosis and treatment for hypertension in Dar es Salaam, Tanzania. Few previous studies in Tanzania have analyzed the modifiable determinants of high BP as well as barriers to diagnosis and treatment of hypertension.

DUCS-HTN is a cohort of adults living in the Ukonga ward of Dar es Salaam who had been registered in the Dar es Salaam Health and Demographic Surveillance System (HDSS) in 2011. Due to the large size of Ukonga, the investigators chose to randomly sample two of the seven neighborhoods that compose Ukonga and then conducted a census of these two randomly selected neighborhoods, Mwembe Madafu and Markazi. The investigators attempted to contact all 4896 HDSS participants who were at least 40 years of age and lived in one of these neighborhoods.

Trained interviewers conducted face-to-face interviews and physical examinations in participants' homes from March to June 2014. Follow-up visits were conducted from April to June 2015.

Among 4896 potentially eligible participants from the HDSS baseline survey, 3604 (74%) were still living at the same address in 2014. Of these, 2290 (64%) enrolled in the DUCS-HTN study. Of the participants enrolled at baseline, 1752 (77%) participated in the follow-up study.

Blood pressure measurements

Trained interviewers measured blood pressure with digital blood pressure monitors (15 Omron M2 and 5 Beurer BM 40 monitors). Standard, large, and extra-large cuff sizes were used according to the size of a participant's arm. Blood pressure was measured three times with at least a 5-minute rest before the first measurement and 3-minute rests between each subsequent measurement. Blood pressure was taken on the left arm with the participant seated and the arm straight at heart level. Usual blood pressure values were calculated as the mean of the second and third readings. If a second visit was conducted, usual blood pressure values were defined as the mean of the second and third readings at both the first and second visits.

Hypertension was defined as SBP≥140 mmHg or DBP≥90 mmHg, or self-reported use of anti-hypertensive medication. Grade I hypertension was defined as SBP of 140 to 159 or DBP of 90 to 99 mmHg; grade II hypertension was defined as SBP of 160 to 179 or DBP of 100 to 109 mmHg; and grade III hypertension was defined as SBP≥180 or DBP≥110 mmHg. Hypertension control was defined as current antihypertensive use and blood pressure of less than 140/90 mmHg. If a participant was found to have grade I or II hypertension, a second visit was scheduled, at least three days later. Those with grade III hypertension at the last reading of the first visit or grade I or II hypertension at the last reading of the second visit were told that they had high blood pressure, advised to see a health professional and were given a referral letter. In addition, a second visit and blood pressure reading was scheduled for a random sample of one-fifth of participants, who were selected for additional blood, urinary, and dietary measurements.

Assessment of covariates

All participants were administered a socio-demographic and lifestyle questionnaire and had their height, weight, and waist and hip circumference measured. Some demographic information (age, sex, neighborhood, religion, and assets used to create a household wealth index) was previously recorded during the HDSS baseline. Information on household health insurance coverage was collected in 2015 as part of routine HDSS updates.

Standard protocols were used to take anthropometric measurements. Participants were weighed with minimal clothing using a digital scale (Seca, Germany) to the nearest 0.1kg and height was measured, with participants not wearing shoes, to the nearest 1cm. Body mass index (BMI) was calculated as the ratio of weight in kilograms to height in meters squared (kg/m2) and categorized according to WHO categories.

The Global Physical Activity Questionnaire (GPAQ) was used to assess physical activity for work, transportation, and leisure. The investigators defined physical inactivity according to WHO guidelines. Number of servings of alcoholic beverages consumed was reported over the past 30 days. The investigators assumed 14 grams of alcohol as a standard drink portion size. A household wealth index was created through a principal component analysis of household characteristics and assets, and was categorized into quintiles. In the follow-up visit, participants were asked about their health over the past year and the reasons for not seeking hypertension care.

A subsample of ~ one fifth of the participants completed a food frequency questionnaire, two 24-hour dietary recalls, a 24-hour urine collection for sodium, creatinine, protein, and potassium, and had capillary total cholesterol and blood glucose measurements taken.

ELIGIBILITY:
Inclusion Criteria:

* Lived in Madafu or Markazi neighborhoods of Ukonga Ward in Tanzania

Exclusion Criteria:

* Pregnant
* Mentally or physically disabled

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: DUCS-HTN is a cohort of adults living in the Ukonga ward of Dar es Salaam who had been registered in the Dar es Salaam Health and Demographic Surveillance System (HDSS) in 2011. Due to the large size of Ukonga, we chose to randomly sample two of the seven neighborhoods that compose Ukonga and then conducted a census of these two randomly selected neighborhoods, Mwembe Madafu and Markazi. We attempted to contact all 4896 HDSS participants who were at least 40 years of age and lived in one of these neighborhoods.
  Trained interviewers conducted face-to-face interviews and physical examinations in participants' homes from March to June 2014. Follow-up visits were conducted from April to June 2015.
  Among 4896 potentially eligible participants from the HDSS baseline survey, 3604 (74%) were still living at the same address in 2014. Of these, 2290 (64%) enrolled in the DUCS-HTN study. Of the participants enrolled at baseline, 1752 (77%) participated in the follow-up study.
Sampling Method: Probability Sample
Enrollment: 2290 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | baseline
  Continuous variable
Visited health professional for hypertension care | 1-year follow-up
  Self report of visiting health professional for hypertension care between baseline and follow-up
Taking antihypertensive medication | 1-year follow-up
  Self report of taking antihypertensive treatment at time of follow-up

SECONDARY OUTCOMES:
Diastolic blood pressure | baseline
Hypertension | baseline
  SBP >=140 or DBP >=90 or using antihypertensive medication